CLINICAL TRIAL: NCT02259972
Title: Investigation of Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of 5 to 800 mg BI 113823 Powder in Bottle (PiB) and Tablet Administered to Healthy Male Volunteers in a Partially Randomised and Double Blinded, Placebo Controlled Phase I Trial. Including Intra-individual Open Comparisons of PiB and Tablet (Fasted and Fed).
Brief Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 113823 Powder in Bottle (PiB) and Tablet in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1272.1
Record Dates: First submitted 2014-10-07; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (3):
- BI 113823 solution (Experimental): single rising doses, dose group 5 twice (fed and fasted)
  Interventions: Drug: BI 113823 solution; Other: High fat, high calorie breakfast
- BI 113823 tablet (Experimental): dose group 5 only
  Interventions: Drug: BI 113823 tablet; Other: High fat, high calorie breakfast
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 113823 solution
  Arms: BI 113823 solution
Drug: BI 113823 tablet
  Arms: BI 113823 tablet
Drug: Placebo
  Arms: Placebo
Other: High fat, high calorie breakfast — only for dose group 5
  Arms: BI 113823 solution; BI 113823 tablet

SUMMARY:
To investigate the safety, tolerability, and pharmacokinetics incl. dose proportionality of BI 113823, as well as the relative bioavailability of PiB vs. tablet and tablet fasted vs. fed (food effect for the tablet).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
2. Age ≥18 and Age ≤45 years
3. BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration
10. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration
11. Participation in another trial with an investigational drug within two months prior to administration or during the trial
12. Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
13. Inability to refrain from smoking on trial days
14. Alcohol abuse (more than 30 g/day)
15. Drug abuse
16. Blood donation (more than 100 mL within four weeks prior to administration)
17. Excessive physical activities (within one week prior to administration)
18. Any laboratory value outside the reference range that is of clinical relevance
19. Inability to comply with dietary regimen of trial site
20. Bradycardia < 50/min, PR interval > 200 ms, QRS interval > 110 ms, QTcB > 450 ms, or QT (uncorrected) > 470 ms or any other relevant ECG findings at screening
21. A history of additional risk factors for Torsades des Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinically significant findings on physical examination | up to 14 days after last drug administration
Number of participants with clinically significant findings in vital signs | up to 14 days after last drug administration
  blood pressure (BP), pulse rate (PR)
Number of participants with clinically significant findings in 12-lead electrocardiogram (ECG) | up to 14 days after last drug administration
  special attention to QRS prolongation
Number of participants with clinically significant findings in laboratory tests | up to 14 days after last drug administration
Number of participants with adverse events | up to 14 days after last drug administration
Assessment of tolerability by investigator on a 4-point scale | up to 14 days after last drug administration

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 72 hours after drug administration
tmax (time from dosing to maximum measured concentration) | up to 72 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 72 hours after drug administration
AUC0-tz (area under the concentration-time curve of metformin in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 72 hours after drug administration
λz (terminal rate constant in plasma) | up to 72 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 72 hours after drug administration
MRToral (mean residence time of the analyte in the body after oral administration) | up to 72 hours after drug administration
CL/F (total/apparent clearance of the analyte in plasma after extravascular administration) | up to 72 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 72 hours after drug administration
Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) | up to 72 hours after drug administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | up to 72 hours after drug administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 72 hours after drug administration